CLINICAL TRIAL: NCT06439953
Title: Impact of Prophylactic Use of Irrisept Irrigation System for Spinal Instrumentation
Brief Title: Irrisept Solution for Instrumented Spine Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2095643
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-06

CONDITIONS: Post-Op Complication; Spine Surgery; Site Infection; Surgical Site Infection; Spinal Instrumentation; Index Spinal Instrumentation; Layer-by-Layer Closure; Locoregional Flap-Based Closure
MeSH Terms: conditions — Postoperative Complications; Surgical Wound Infection | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Irrisept Irrigation (Experimental): Patients scheduled to undergo spinal instrumentation will receive intra-operative Irrisept irrigation.
  Interventions: Device: Chlorhexidine gluconate solution
- Vancomycin-saline Irrigation (Active Comparator): Patients scheduled to undergo spinal instrumentation will receive intra-operative irrigation using vancomycin-saline irrigation.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Device: Chlorhexidine gluconate solution — Evaluating the prophylactic use of Irrisept irrigation alone
  Other Names: Irrisept irrigation
  Arms: Irrisept Irrigation
Drug: Vancomycin — Evaluating the use of versus vancomycin-saline irrigation with or without topical vancomycin
  Other Names: Vancomycin-saline
  Arms: Vancomycin-saline Irrigation

SUMMARY:
Various spine surgeons perform wound irrigation using saline mixed with vancomycin, relying on mechanical debridement of non-viable tissue, physical disruption of biofilm, and bacteriostatic effect against gram positive flora. When used as a powder, topical application of vancomycin has demonstrated increased risk of symptomatic seroma formation, which is an adverse outcome that often requires bedside or intra-operative aspiration. Broad-spectrum antiseptic agents, such as Irrisept, offer bacteriocidal properties to eliminate hardware inoculation, thereby minimizing the risk of deep space infection, while obviating the risk of seroma development.

DETAILED DESCRIPTION:
Spinal instrumentation remains the standard of care in the treatment of various traumatic, oncologic, and degenerative spinal pathologies, often requiring the implantation of hardware to stabilize the bony column. In the setting of an aging patient population and expanding indications for instrumentation in younger patients, the number of spinal operations performed has risen substantially within the past decade. Although these procedures have proven to enhance patient quality of life, spinal instrumentation is not without post-operative complication, most notable of which are surgical site infection, seroma formation, and wound breakdown. Such complications can result in notable negative sequelae. Recurrent seroma may compress underlying neurologic structures or increase pressure along the incision, thereby precipitating wound dehiscence and inoculation of the surgical site with pathogenic organisms. Deep space infections often result in prolonged hospitalization, long-term suppressive antibiotic therapy, hardware removal, and permanent disability, which increases cost burden at the patient and hospital level. As such, preventative strategies to reduce the rate of complications following spinal instrumentation remain paramount. Within recent years, attention has turned to various irrigation methods to terminally sterilize prosthetic devices and wound beds, thereby minimizing bacterial colonization and biofilm formation that would otherwise predispose infection.

Irrisept (Irrimax Corporation, Gainesville, Florida) is a solution comprised of 0.05% chlorhexidine gluconate in 99.95% sterile water administered through a proprietary, low-pressure lavage mechanism that has demonstrated efficacy as a bacteriocidal agent in orthopedic hip and knee arthroplasty procedures. Whereas other antiseptic irrigation solutions, such as vancomycin-saline lavage, are routinely used to prevent surgical site infection, relative inertness against gram negative organisms and potential predisposition toward seroma formation render them non-ideal for use in spine surgery. Despite the utility of dilute chlorhexidine gluconate as a prophylactic irrigant, there exist gaps in knowledge with regard to the efficacy of Irrisept to prevent post-operative complications following spinal instrumentation. The central hypothesis of this proposal is that prophylactic use of Irrisept irrigation will result in fewer surgical site infections, clinically significant seromas, and gram negative or atypical infections when compared to standard of care irrigation (vancomycin-saline solution with or without topical vancomycin powder).

Proposed is a prospective, randomized controlled trial comparing rates of post-operative complications following use of Irrisept irrigation alone versus vancomycin-saline lavage with or without topical vancomycin powder (standard of care) in patients aged 18 years or older who undergo posterior cervical, thoracic, lumbar, and/or sacral spinal instrumentation for various indications (deformity, malignancy, degenerative pathology, and trauma) at Rhode Island Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18+ years old
* Indications: deformity, oncologic, degenerative, trauma
* Standard layer-by-layer closure
* Locoregional flap-based closure

Exclusion Criteria:

* Acute/chronic open wounds (spine or non-spine)
* On-going non-spinal infection within 30 days of index operation
* Concurrent antibiotic use (for spine or non-spine infections)
* History of prior spinal infection
* Allergy to vancomycin or chlorhexidine
* Suspicion for osteomyelitis
* Other surgery within 90 days post-operatively fromm index
* Concurrent enrollment in other trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of surgical site infection | 90 days post-operatively
  Development of infection after index spinal instrumentation

SECONDARY OUTCOMES:
Mortality | 12 months post-operatively
  Capture mortality rates after index spinal instrumentation
Duration of index hospitalization | 12 months post-operatively
  Capture duration of index hospitalization after index spinal instrumentation
Occurrence of 30-day readmission | 30 days post-operatively
  Capture 30-day readmission rates after index spinal instrumentation
Occurrence of wound dehiscence | 12 months post-operatively
  Capture all incidences of wound dehiscence after index spinal instrumentation
Time to closed suction drain removal | 12 months post-operatively
  Capture the time interval to closed suction drain removal after index spinal instrumentation
Presence of atypical micro-organisms on wound fluid laboratory culture | 12 months post-operatively
  Capture the presence of atypical micro-organisms after index spinal instrumentation
Cost of spine surgery care from surgery to 12-month post-operative follow up | 12 months post-operatively
  Consider associated total costs of spinal instrumentation after index spinal instrumentation by comparing total surgical costs and post-surgical outcome expenses of those with and without Irrisept irrigation use

CONTACTS AND LOCATIONS:
Overall Officials: Jared S. Fridley, MD, Principal Investigator — Rhode Island Hospital; Albert S. Woo, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deyo RA, Mirza SK, Martin BI, Kreuter W, Goodman DC, Jarvik JG. Trends, major medical complications, and charges associated with surgery for lumbar spinal stenosis in older adults. JAMA. 2010 Apr 7;303(13):1259-65. doi: 10.1001/jama.2010.338. PMID 20371784
- [Background] Martin BI, Mirza SK, Spina N, Spiker WR, Lawrence B, Brodke DS. Trends in Lumbar Fusion Procedure Rates and Associated Hospital Costs for Degenerative Spinal Diseases in the United States, 2004 to 2015. Spine (Phila Pa 1976). 2019 Mar 1;44(5):369-376. doi: 10.1097/BRS.0000000000002822. PMID 30074971
- [Background] Jain NK, Dao K, Ortiz AO. Radiologic evaluation and management of postoperative spine paraspinal fluid collections. Neuroimaging Clin N Am. 2014 May;24(2):375-89. doi: 10.1016/j.nic.2014.01.001. PMID 24792615
- [Background] Blumberg TJ, Woelber E, Bellabarba C, Bransford R, Spina N. Predictors of increased cost and length of stay in the treatment of postoperative spine surgical site infection. Spine J. 2018 Feb;18(2):300-306. doi: 10.1016/j.spinee.2017.07.173. Epub 2017 Jul 21. PMID 28739477
- [Background] de Lissovoy G, Fraeman K, Hutchins V, Murphy D, Song D, Vaughn BB. Surgical site infection: incidence and impact on hospital utilization and treatment costs. Am J Infect Control. 2009 Jun;37(5):387-397. doi: 10.1016/j.ajic.2008.12.010. Epub 2009 Apr 23. PMID 19398246
- [Background] Torres KA, Konrade E, White J, Tavares Junior MCM, Bunch JT, Burton D, Jackson RS, Birlingmair J, Carlson BB. Irrigation techniques used in spine surgery for surgical site infection prophylaxis: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2022 Aug 26;23(1):813. doi: 10.1186/s12891-022-05763-2. PMID 36008858
- [Background] Yao R, Tan T, Tee JW, Street J. Prophylaxis of surgical site infection in adult spine surgery: A systematic review. J Clin Neurosci. 2018 Jun;52:5-25. doi: 10.1016/j.jocn.2018.03.023. Epub 2018 Mar 30. PMID 29609860
- [Background] Kapadia BH, Zhou PL, Jauregui JJ, Mont MA. Does Preadmission Cutaneous Chlorhexidine Preparation Reduce Surgical Site Infections After Total Knee Arthroplasty? Clin Orthop Relat Res. 2016 Jul;474(7):1592-8. doi: 10.1007/s11999-016-4767-6. PMID 26956247
- [Background] Johnson AJ, Kapadia BH, Daley JA, Molina CB, Mont MA. Chlorhexidine reduces infections in knee arthroplasty. J Knee Surg. 2013 Jun;26(3):213-8. doi: 10.1055/s-0032-1329232. Epub 2012 Nov 12. PMID 23288739
- [Background] Lung BE, Le R, Callan K, McLellan M, Issagholian L, Yi J, McMaster WC, Yang S, So DH. Chlorhexidine gluconate lavage during total joint arthroplasty may improve wound healing compared to dilute betadine. J Exp Orthop. 2022 Jul 10;9(1):67. doi: 10.1186/s40634-022-00503-w. PMID 35819733
- [Background] Ghobrial GM, Cadotte DW, Williams K Jr, Fehlings MG, Harrop JS. Complications from the use of intrawound vancomycin in lumbar spinal surgery: a systematic review. Neurosurg Focus. 2015 Oct;39(4):E11. doi: 10.3171/2015.7.FOCUS15258. PMID 26424335
- [Background] Youssef JA, Orndorff DG, Scott MA, Ebner RE, Knewitz AP. Sterile Seroma Resulting from Multilevel XLIF Procedure as Possible Adverse Effect of Prophylactic Vancomycin Powder: A Case Report. Evid Based Spine Care J. 2014 Oct;5(2):127-33. doi: 10.1055/s-0034-1386754. PMID 25364326
- [Background] Mallet C, Meissburger V, Caseris M, Happiette A, Chinnappa J, Bonacorsi S, Simon AL, Ilharreborde B. Does the use of intrawound povidone-iodine irrigation and local vancomycin powder impact surgical site infection rate in adolescent idiopathic scoliosis surgery? Eur Spine J. 2022 Nov;31(11):3020-3028. doi: 10.1007/s00586-022-07340-6. Epub 2022 Aug 1. PMID 35913622
- [Background] Schroeder JE, Girardi FP, Sandhu H, Weinstein J, Cammisa FP, Sama A. The use of local vancomycin powder in degenerative spine surgery. Eur Spine J. 2016 Apr;25(4):1029-33. doi: 10.1007/s00586-015-4119-3. Epub 2015 Aug 7. PMID 26249032
- [Background] Lemans JVC, Oner FC, Wijdicks SPJ, Ekkelenkamp MB, Vogely HC, Kruyt MC. The efficacy of intrawound vancomycin powder and povidone-iodine irrigation to prevent surgical site infections in complex instrumented spine surgery. Spine J. 2019 Oct;19(10):1648-1656. doi: 10.1016/j.spinee.2019.05.592. Epub 2019 May 31. PMID 31158503
- [Background] Cohen LE, Fullerton N, Mundy LR, Weinstein AL, Fu KM, Ketner JJ, Hartl R, Spector JA. Optimizing Successful Outcomes in Complex Spine Reconstruction Using Local Muscle Flaps. Plast Reconstr Surg. 2016 Jan;137(1):295-301. doi: 10.1097/PRS.0000000000001875. PMID 26710033
- [Background] Rinkinen JR, Weitzman RE, Clain JB, Lans J, Shin JH, Eberlin KR. Locoregional Flap Closure for High-risk Multilevel Spine Surgery. Plast Reconstr Surg Glob Open. 2020 Apr 21;8(4):e2751. doi: 10.1097/GOX.0000000000002751. eCollection 2020 Apr. PMID 32440420
- [Background] Hochberg J, Ardenghy M, Yuen J, Gonzalez-Cruz R, Miura Y, Conrado RM, Pait TG. Muscle and musculocutaneous flap coverage of exposed spinal fusion devices. Plast Reconstr Surg. 1998 Aug;102(2):385-9; discussion 390-2. doi: 10.1097/00006534-199808000-00013. PMID 9703074